CLINICAL TRIAL: NCT04358770
Title: Single Exposure Bioequivalence Study to Evaluate the Vasoconstriction Activity of Topically Applied Cloderm® (Clocortolone Pivalate) 0.1% Cream and Clocortolone Pivalate 0.1% Cream (Taro Pharmaceuticals) in Healthy Male and Female Volunteers With Normal Skin Under Occlusive Conditions.
Brief Title: Bio-equivalence Vasoconstriction Activity Study for Topically Applied Clocortolone Pivalate 0.1% Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Collaborators: WAYCro (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CLPC-1801
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Bioequivalence Study
MeSH Terms: interventions — clocortolone pivalate; clocortolone

STUDY DESIGN:
Intervention Model Description: single-exposure, open-label, vasoconstriction response study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (Experimental): Clocortolone Pivalate Cream, 0.1%
  Interventions: Drug: Clocortolone Pivalate
- Reference (Active Comparator): Cloderm® (clocortolone pivalate) Cream, 0.1%
  Interventions: Drug: Clocortolone Pivalate

INTERVENTIONS:
Drug: Clocortolone Pivalate — Cream, 0.1%
  Other Names: Clocortolone

SUMMARY:
To compare pharmacodynamic vasoconstriction response profile of Clocortolone Pivalate 0.1% Cream and Cloderm® (Clocortolone Pivalate) 0.1% Cream in normal skin of healthy male and female adults

ELIGIBILITY:
Inclusion Criteria:

* Normal or clinically insignificant dermatological history the Screening visit and Day 1dosing;

Exclusion Criteria:

* Female subjects who were pregnant, nursing, or planning to become pregnant during study participation;
* History of hypersensitivity to the study products or any topical or systemic corticosteroids;

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
AUEC0-24 (area under the effect curve) | 24 hours
  value for the blanching intensity vs. time profile

CONTACTS AND LOCATIONS:
Locations (1):
- WayCro, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No